CLINICAL TRIAL: NCT04600375
Title: Evaluating the Effect of a Written Action Plan on Comfort and Understanding of Hidradenitis Suppurativa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 261683
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Results first posted 2022-04-06 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-02

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbal Consultation, then Written Action Plan (Other): CONTROL GROUP
  1. Survey A
  2. Routine clinic visit
  3. Verbal consultation only
  4. Survey B
  5. Verbal consultation AND Written Action Plan
  6. Survey C
  Interventions: Behavioral: Verbal consultation; Behavioral: Written Action Plan
- Experimental: Written Action Plan (Experimental): INTERVENTION GROUP
  1. Survey A
  2. Routine clinic visit
  3. Verbal consultation AND Written Action Plan
  4. Survey C
  Interventions: Behavioral: Written Action Plan

INTERVENTIONS:
Behavioral: Verbal consultation — Verbal consultation only without written information before receiving written action plan
  Arms: Verbal Consultation, then Written Action Plan
Behavioral: Written Action Plan — Written handout of treatment plan and disease management strategies

SUMMARY:
This study is being conducted to evaluate if a written action plan for hidradenitis suppurativa (HS) will help patients with hidradenitis suppurativa gain a better understanding of the condition and how to manage the condition on a daily basis compared to a routine verbal consultation.

ELIGIBILITY:
Inclusion Criteria:

* This study will only enroll subjects between the ages of 18-years and 89-years of age.
* Diagnosis of HS by a board-certified dermatologist
* Able to read and comprehend study materials
* No prior exposure to written HS action plans

Exclusion Criteria:

* Those who do not fit the inclusion criteria

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Y Shi, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Thompson AM, Fernandez JM, Shih T, Hamzavi I, Hsiao JL, Shi VY. Improving hidradenitis suppurativa patient education using written action plan: a randomized controlled trial. J Dermatolog Treat. 2022 Aug;33(5):2677-2679. doi: 10.1080/09546634.2021.1970707. Epub 2021 Sep 27. PMID 34579620

RESULTS

PARTICIPANT FLOW:
Groups:
- Verbal Consultation, Then Written Action Plan: CONTROL GROUP
  1. Survey A
  2. Routine clinic visit
  3. Verbal consultation only
  4. Survey B
  5. Verbal consultation AND Written Action Plan
  6. Survey C
  Verbal consultation: Verbal consultation only without written information before receiving written action plan
  Written Action Plan: Written handout of treatment plan and disease management strategies
- Experimental: Written Action Plan: INTERVENTION GROUP
  1. Survey A
  2. Routine clinic visit
  3. Verbal consultation AND Written Action Plan
  4. Survey C
  Written Action Plan: Written handout of treatment plan and disease management strategies
Period: Overall Study
Arm/Group | Verbal Consultation, Then Written Action Plan | Experimental: Written Action Plan
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verbal Consultation, Then Written Action Plan | Experimental: Written Action Plan | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (8.6) | 34.2 (11.9) | 33.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 0 | 5 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Visits to High-cost Care Settings [ Time Frame: 1.5 Months ]
Description: Number of visits to ER, urgent care, or hospitalizations because of HS
Time Frame: Through study completion, an average of 1.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Verbal Consultation, Then Written Action Plan | Experimental: Written Action Plan
Number analyzed (Participants) | 12 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1.5 months.
Description: Not different from clinicaltrials.gov definition
Arm/Group | Verbal Consultation, Then Written Action Plan | Experimental: Written Action Plan
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT04600375/Prot_SAP_000.pdf